CLINICAL TRIAL: NCT07239908
Title: Resuscitation Enhancement to Avoid Rearrest Through Evidence-based Strategies in Prehospital Post-resuscitation Care
Acronym: RE-ARREST
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Sattha Riyapan, Assistant professor, Siriraj Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 801/2568(IRB4)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
Keywords: Post cardiac arrest care; Out-of-hospital cardiac arrest; Prehospital care
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Prehospital post cardiac arrest care protocol for advanced life support ambulance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): Conventional post cardiac arrest care by ALS unit in Bangkok Thailand
- Prehospital post cardiac arrest care protocol (Experimental): Prehospital post cardiac arrest care protocol
  Interventions: Drug: Prehospital post cardiac arrest care protocol

INTERVENTIONS:
Drug: Prehospital post cardiac arrest care protocol — Prehospital post cardiac arrest care including:
  1. Fluid assessment and resuscitation in prehospital phase
  2. Early vasopressor in prehospital phase
  3. Regular monitoriny end-tidal CO2 in prehospital phase
  Arms: Prehospital post cardiac arrest care protocol

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) remains a leading global emergency condition with low survival to hospital discharge despite advances in cardiopulmonary resuscitation. Return of spontaneous circulation (ROSC) rates have improved; however, 30-50% of patients experience rearrest after ROSC, which is associated with significantly reduced survival. Preventable physiologic factors related to prehospital care - including hypoxia, hypotension, and hyperventilation - are frequently identified prior to rearrest. Evidence-based post-ROSC clinical bundles exist mainly for in-hospital settings, while structured prehospital post-resuscitation care protocols are limited, particularly in resource-constrained environments.

The RE-ARREST project aims to develop, implement, and evaluate an evidence-based prehospital post-resuscitation care protocol designed for paramedic-led Emergency Medical Services. The intervention includes structured monitoring, tailored oxygenation and ventilation targets, vasopressor use criteria (norepinephrine), fluid management decision support, teamwork communication, and operational training workshops using simulation.

This is a quasi-experimental pre-post interventional study conducted at the Siriraj Emergency Medical Service (SiEMS), Thailand. The study compares outcomes from retrospective pre-implementation cases with prospective post-implementation cases, including both patient-centered outcomes and provider compliance. Adult OHCA patients with ROSC achieved prehospital and transported to Siriraj Hospital are eligible. The estimated sample size is 318 participants (pre-intervention 212; post-intervention 106) over two years.

The primary outcome is the incidence of rearrest within 1 hour after ROSC during prehospital care and initial emergency department management. Secondary outcomes include protocol compliance, survival-to-admission, and survival-to-hospital-discharge. The protocol emphasizes feasibility, safety, and replicability to inform scalable EMS clinical practice guidelines.

This research is expected to provide novel evidence on targeted prehospital post-ROSC care and has the potential to reduce rearrest, improve neurologically favorable survival, and strengthen EMS system quality improvement efforts in Thailand and other low-to-middle-resource settings.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients who has out-of-hospital cardiac arrest
2. patients who has return of spontaneous circulation after OHCA

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Rearrest rate | From return of spontaneous circulation to first 1 hour in emergency room
  patient who has return of spontaneous circulation and then has no pulse again

SECONDARY OUTCOMES:
Survival to dischrage | 30 days after admission
  patient who survival after admit to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sattha Riyapan, MD MPH, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Vos IA, Lucassen FG, Bens BWJ, Dercksen B, Postma R, Jorna EMF, Ter Maaten JC, Struys MMRF, Ter Avest E. Pre-hospital care after return of spontaneous circulation: Are we achieving our targets? Resusc Plus. 2024 Jun 21;19:100691. doi: 10.1016/j.resplu.2024.100691. eCollection 2024 Sep. PMID 39006133
- [Background] Dillon DG, Montoy JCC, Bosson N, Toy J, Kidane S, Ballard DW, Gausche-Hill M, Donofrio-Odmann J, Schlesinger SA, Staats K, Kazan C, Morr B, Thompson K, Mackey K, Brown J, Menegazzi JJ; California Resuscitation Outcomes Consortium. Rationale and development of a prehospital goal-directed bundle of care to prevent rearrest after return of spontaneous circulation. J Am Coll Emerg Physicians Open. 2024 Nov 5;5(6):e13321. doi: 10.1002/emp2.13321. eCollection 2024 Dec. PMID 39503017
- [Background] Toy J, Tolles J, Bosson N, Hauck A, Abramson T, Sanko S, Kazan C, Eckstein M, Gausche-Hill M, Schlesinger SA. Association between a Post-Resuscitation Care Bundle and the Odds of Field Rearrest after Successful Resuscitation from Out-of-Hospital Cardiac Arrest: A Pre/Post Study. Prehosp Emerg Care. 2024;28(1):98-106. doi: 10.1080/10903127.2023.2172633. Epub 2023 Feb 13. PMID 36692410
- [Background] Smida T, Price BS, Mizener A, Crowe RP, Bardes JM. Prehospital Post-Resuscitation Vital Sign Phenotypes are Associated with Outcomes Following Out-of-Hospital Cardiac Arrest. Prehosp Emerg Care. 2025;29(2):138-145. doi: 10.1080/10903127.2024.2386445. Epub 2024 Aug 15. PMID 39088816
- [Background] Smida T, Menegazzi JJ, Crowe RP, Weiss LS, Salcido DD. Association of prehospital hypotension depth and dose with survival following out-of-hospital cardiac arrest. Resuscitation. 2022 Nov;180:99-107. doi: 10.1016/j.resuscitation.2022.09.018. Epub 2022 Sep 30. PMID 36191809
- [Background] Salcido DD, Sundermann ML, Koller AC, Menegazzi JJ. Incidence and outcomes of rearrest following out-of-hospital cardiac arrest. Resuscitation. 2015 Jan;86:19-24. doi: 10.1016/j.resuscitation.2014.10.011. Epub 2014 Oct 23. PMID 25447433
- [Background] Salcido DD, Stephenson AM, Condle JP, Callaway CW, Menegazzi JJ. Incidence of rearrest after return of spontaneous circulation in out-of-hospital cardiac arrest. Prehosp Emerg Care. 2010 Oct-Dec;14(4):413-8. doi: 10.3109/10903127.2010.497902. PMID 20809686
- [Background] Lerner EB, O'Connell M, Pirrallo RG. Rearrest after prehospital resuscitation. Prehosp Emerg Care. 2011 Jan-Mar;15(1):50-4. doi: 10.3109/10903127.2010.519820. Epub 2010 Nov 5. PMID 21054177
- [Background] Chestnut JM, Kuklinski AA, Stephens SW, Wang HE. Cardiovascular collapse after return of spontaneous circulation in human out-of-hospital cardiopulmonary arrest. Emerg Med J. 2012 Feb;29(2):129-32. doi: 10.1136/emj.2010.108340. Epub 2011 Feb 18. PMID 21335581
- [Background] Woo JH, Cho JS, Lee CA, Kim GW, Kim YJ, Moon HJ, Park YJ, Lee KM, Jeong WJ, Choi IK, Choi HJ, Choi HJ. Survival and Rearrest in out-of-Hospital Cardiac Arrest Patients with Prehospital Return of Spontaneous Circulation: A Prospective Multi-Regional Observational Study. Prehosp Emerg Care. 2021 Jan-Feb;25(1):59-66. doi: 10.1080/10903127.2020.1733716. Epub 2020 Mar 20. PMID 32091295
- [Background] Berdowski J, Berg RA, Tijssen JG, Koster RW. Global incidences of out-of-hospital cardiac arrest and survival rates: Systematic review of 67 prospective studies. Resuscitation. 2010 Nov;81(11):1479-87. doi: 10.1016/j.resuscitation.2010.08.006. Epub 2010 Sep 9. PMID 20828914